CLINICAL TRIAL: NCT01013610
Title: A Double-Blind, Randomized, Placebo-Controlled, Multiple, Escalating Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LNK 754 in Elderly Volunteers and in Subjects With Mild Alzheimer's Disease
Brief Title: An Escalating Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LNK 754 in Elderly Volunteers and in Subjects With Mild Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Link Medicine Corporation (Industry)
Responsible Party: Scott Young, Chief Operating Officer, Link Medicine Corporation
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: LNK754-0902-1AB
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Mild Alzheimer's Disease
Keywords: Healthy Elderly Volunteers
MeSH Terms: interventions — LNK-754

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiple Dose (Active Comparator)
  Interventions: Drug: LNK-754
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LNK-754 — Escalating dose
  Arms: Multiple Dose
Drug: Placebo — Escalating dose
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability, multiple dose plasma pharmacokinetics (PK) of LNK-754 in male and female elderly volunteers after dosing with LNK-754 for 7 days and in subjects with mild Alzheimer's Disease after dosing with LNK-754 for 28 days.

ELIGIBILITY:
Inclusion Criteria:

Part A and Part B:

1. Males or females aged 60 years or older. Females must be surgically sterilized or postmenopausal for at least two years. Males must be actively practicing double-barrier contraception (condom plus spermicide), unless they have had a vasectomy, or their partner(s) meet the above criteria for females.
2. Voluntarily consent to participate in this study and provide written informed consent prior to start of any study-specific procedures.
3. Be prepared to adhere to the protocol requirements and be willing and able to remain in the study unit for the entire duration of the confinement period. They must also be willing to return for the End-of-Study Visit one week after the last dosing.

   Part A only:
4. Subjects must be generally healthy, but may be enrolled with a stable, chronic illness, if it is well controlled and does not interfere with the primary objective of the study. Subjects may be included with clinical deviations from normal limits in medical history, physical examination, vital sign measurements, ECG, or laboratory test results that are associated with stable, well controlled chronic illness. Subjects with concomitant diseases or using concomitant medication will be allowed to participate provided a stable condition and stable treatment for 1 month (30 days) prior to administration of the first dose of study medication. Inclusion of each subject will be reviewed with the Link Medical Monitor prior to enrollment in the trial.

   Part B only:
5. Subjects with Mild Alzheimer's Disease, as defined by DSM-IV.
6. Subjects with a score of ≥ 18-26 on the Mini-Mental State Examination (MMSE).
7. Subjects with a Clinical Dementia Rating (CDR) total score of 0.5 or 1.0 (possible or mild dementia).
8. Subjects with a Rosen-Modified Hachinski Ischemic score of ≤ 4.

Exclusion Criteria:

Part A and Part B:

1. Any significant unstable or uncontrolled cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease, as determined by medical history, physical examination or laboratory tests.
2. Subjects who have positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
3. Subjects who have received any experimental drugs or devices within 30 days prior to dosing or who wish to receive any experimental drug within 30 days after completing the study.
4. Subjects unable to understand the protocol requirements, instructions and study related restrictions, the nature, scope and possible consequences of the clinical study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety assessments to include pharmacokinetics, and adverse events | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riesenberg, MD, Principal Investigator — Atlanta Center for Medical Research; Abel Murillo, MD, Principal Investigator — Elite Research Institute; Craig T. Curtis, MD, Principal Investigator — Compass Research; Kyle Patrick, D.O., Principal Investigator — Dedicated Phase I; Maxwell Axler, MD, Principal Investigator — Clinical Trial Network; Ricky S. Mofsen, D.O., Principal Investigator — St. Louis Clinical Trials, LC; Armen Goenjian, MD, Principal Investigator — Collaborative Neuroscience Network
Locations (7):
- United States (7):
  - Dedicated Phase I, Phoenix, Arizona
  - Collaborative Neuroscience Network, Long Beach, California
  - Elite Research Insitute, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - Clinical Trial Network, Houston, Texas